CLINICAL TRIAL: NCT04878419
Title: Acceptability of a Virtual Educational Intervention Targeted Towards Improving Diabetes Self- Efficacy and Glycemic Control in Adolescents and Young Adults With Type 1 Diabetes Mellitus (T1DM): a Pilot Study
Brief Title: Acceptability of Virtual Educational Intervention for Adolescents and Young Adults With Type 1 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Jamie Wood, Pediatric Endocrinologist, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY20210264
Record Dates: First submitted 2021-04-28; First posted 2021-05-07 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Self efficacy; Virtual; Education; Adolescents; Young adults
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Educational Intervention (Experimental): Virtual Educational Intervention
  Interventions: Other: Virtual Educational Program

INTERVENTIONS:
Other: Virtual Educational Program — Multiple virtual interactive sessions to provide education/knowledge about Type 1 Diabetes Mellitus care

SUMMARY:
In this pilot study, study investigators aim to evaluate the acceptability and feasibility of a 3-month interactive virtual educational program, designed on principles of self-efficacy, reviewing aspects of Diabetes Mellitus care in adolescents and young adults with Type 1 Diabetes Mellitus (T1DM). Secondarily, investigators also aim to evaluate the effect of the educational program on participants subjective diabetes self-efficacy, diabetes related knowledge, diabetes distress as well as glycemic control.

Population size:

Fifteen (15) patients will be recruited and enrolled in this study.

Study Design: This is a pilot acceptability and feasibility study with a prospective design to evaluate the effect of the educational intervention on multiple endpoints.

Study Duration:

Participants will complete educational intervention over duration of 3 months after which their glycemic control data will be retrieved from the first clinic visit post intervention (within 5 months of completion of the intervention). Hence, The overall study duration is approximately >3 to 9 months.

DETAILED DESCRIPTION:
Background/Rationale:

The landmark study Diabetes Control and Complications Trial (DCCT, 1982-1993) conclusively proved that intensive glycemic control causes a reduction in the early stages of all microvascular complications of Type 1 Diabetes Mellitus. The durability of the impact of intensive glycemic control in reducing long term microvascular as well as macro vascular complications of T1DM was further endorsed by the observational follow up study 'Epidemiology of Diabetes Interventions and Complications (EDIC). (1)

Intensive glycemic control has since become the primary clinical goal to ensure a healthy, long life for patients with T1DM. In clinical practice, this is truly a challenge. Particularly in pediatric patients, metabolic control worsens during adolescence in both sexes. (2) Physiologic increase in insulin resistance during puberty partly plays a role, but research has shown that psychosocial factors like family functioning, coping skills, depression/anxiety contribute to metabolic control in adolescence. (3,4) Unfortunately, this worsening of metabolic control continues into young adulthood. Glycemic control substantially declines amongst T1D patients in the age range for transition to adult care, with mean HbA1C at its peak of 9.2% at age 19 years after which the glycemic control gradually improves. (5) Of note, between the ages 18-25 years of age, only 14% of patients were shown to meet American Diabetes Association(ADA) HbA1c targets from the updated data from the T1D Exchange Clinic Registry. (5)

T1DM is a chronic lifelong illness that requires self-management on a daily basis. Despite technological leaps in the insulin delivery and blood glucose monitoring devices, self-management remains vital to diabetes mellitus care. Undoubtedly, closed loop systems have taken away the need for frequent Self-Monitoring of Blood Glucose and insulin dose administrations and adjustments, this technology is still fairly new, not universally available, is not personally preferred universally and continues to require awareness of the technological issues and participation in other aspects of Diabetes Mellitus (DM) self-care like diet and exercise.

This self-management role transitions from parent-dominant to shared management to adolescent dominant management over the course of adolescence period. (6) This age group is of particular interest for self-efficacy enhancement studies as the adolescents will soon transition to adulthood and more or less independent self-care. Self- efficacy is one's beliefs about ability to achieve a goal. Metabolic control is affected by perceived self-efficacy to conduct self-care. (7) Self-efficacy beliefs are influenced by mastery, imaginal, vicarious experiences as well as physiological states and social persuasion. (8) Cultivation of positive self-efficacy is very important as it not only influences task performance but also plays a role in coping. (8)

Strategies to improve glycemic control remains an area of interest for clinicians and researchers. In a meta-analysis of ten randomized control trials, Winkley et al concluded that psychological treatments can slightly improve glycemic control in children. (9) Other studies have shown that adherence to treatment regimen is linked to better glycemic control. (10) Literature is rampant with adherence promoting behavioral interventions to positively affect the diabetes self-management. Some examples include motivational/solution-focused group intervention (11), coping skills training (12), family-focused teamwork (TW) intervention (13), diabetes personal trainer" intervention, consisting of self-monitoring, goal-setting, and problem-solving sessions with trained nonprofessionals (14). Meta-analysis of fifteen (randomized control trials (RCTs) that employed adherence promoting behavioral interventions concluded that there is only a modest improvement in glycemic control with significant variability between different interventions. (15)

Unfortunately, most of these interventions are costly, time consuming and not practical for long term maintenance and employment in a clinical setting. Interventions that keep in consideration the concept of reach, efficacy, adoption, implementation, maintenance (RE-AIM) are required. (16)

To tackle these issues, investigators plan to study virtual interventions employing telehealth services. Telehealth videoconferencing has the potential to improve care in pediatric diabetes patients by increasing visits. (17) Studies have shown that patients' glycemic control remained stable and there was no increase in Diabetic Ketoacidosis (DKA), Emergency Department (ED) or hospital visits and satisfaction was equal to in-person visits with telehealth. (18) Virtual access is more stream- lined, overcomes the challenge of time and resources needed on part of patient. Particularly, during the uncertain times of the Coronavirus disease-19 (COVID-19) pandemic, virtual programs can serve a vital role. The study findings can be used to construct a virtual structured transition of care program for youth with Type 1 Diabetes Mellitus which is more accessible and time-flexible for patient needs.

Study Objectives:

1. To evaluate the acceptability and feasibility of a 3-month interactive virtual educational program, designed on principles of self-efficacy, reviewing aspects of Diabetes Mellitus care in adolescents and young adults with Type 1 Diabetes Mellitus.
2. To evaluate the effect of the educational program on participants subjective diabetes self-efficacy, diabetes related knowledge, diabetes distress as well as glycemic control.
3. To evaluate the effect of outcome expectation on degree of change in participants subjective diabetes self-efficacy, diabetes related knowledge, diabetes distress as well as glycemic control after the educational intervention.
4. To evaluate the association of childhood opportunity index with the impact of the educational intervention

Study Hypotheses:

* Investigators hypothesize that the participants will have improvement in their subjective diabetes self-efficacy, diabetes knowledge scores, diabetes distress as well as their glycemic control (measured by percent change in HbA1C and Time in Range data) post-completion of intervention.
* Investigator also hypothesize that participants with positive outcome expectation for the virtual education program and with a higher childhood opportunity score will have greater improvement in their subjective diabetes self- efficacy, diabetes related distress, diabetes knowledge scores and glycemic control post intervention.

Study Design:

This is a pilot acceptability and feasibility study with a prospective design to evaluate the effect of the educational intervention on multiple endpoints.The overall study duration is approximately >3 to 9 months.

Pre-Intervention Procedures:

The following surveys will be administered to the participants at the pre-intervention encounter:

1. A baseline survey about patient's characteristics and diabetes management data.
2. Diabetes Self Efficacy survey
3. Diabetes related Distress survey
4. Diabetes Knowledge survey
5. Survey for Outcome expectation for the intervention

Glycemic control data (HBA1C and Time in Range) will be retrieved from the patient's medical chart from the clinic visit prior to consenting for the study.

Intervention Procedures:

Weekly virtual and interactive educational sessions will be administered by the PI. There are total 11 sessions. Each session is about 15-20 minutes. These sessions will be administered through secure tele-health media Doxy.me. At the end of each module, feedback surveys will be administered.

Broadly, the educational sessions will cover topics including Type 1 Diabetes pathophysiology, management of T1DM and complications of Hypoglycemia and Hyperglycemia, Types of Insulin, available Diabetes technology and utilizing blood glucose data for T1DM management, Sick day management, diabetes related complications, practical life issues during transition to adulthood including insurance, medications and supplies management, driving, dating and impact of drinking and drugs on T1DM management. These modules will also cover anticipated issues during transition to college or to workplace and guidance to mitigate the issues.

Post-Intervention Procedures:

At the completion of the entire 3 month educational program, following surveys will be administered.

1. Feedback survey for the entire educational program.
2. Diabetes Self Efficacy survey
3. Diabetes related Distress survey
4. Diabetes Knowledge survey

Glycemic control data (HBA1C and Time in Range) will be retrieved from the patient's medical chart from the 1st clinic visit after completion of the entire educational program ( within five months of completion of the intervention).

ELIGIBILITY:
Inclusion Criteria:

* Age range: from 16 years to 21 years of age
* Type 1 Diabetes Mellitus (Anti-body positive) for at least one year
* Suboptimal glycemic control (HBA1C > 8.5%) in the last 6 months
* Patients on insulin regimen involving multiple daily subcutaneous insulin injections (basal- bolus regimen) or insulin pumps (excluding hybrid close loop pumps)

Exclusion Criteria:

* Non-English-Speaking patients
* Patients on insulin regimen involving mixed insulin with twice daily injections
* Patients who are planning to undergo any change in their insulin delivering technology or glucose monitoring device during the study time period i.e. planning initiation or discontinuation of pump or Continuous Glucose Meter.
* Patients who received new onset DM teaching at another institution and transferred care from other institutions later in their disease course.
* Individuals with other chronic medical conditions or underlying mental health conditions like eating disorders, schizophrenia or severe depression or inability to care for themselves in activities of daily living (ADLs), or impaired ability to participate in the research in the discretion of their primary diabetes provider.
* Patients lacking accessibility of a virtual platform for the intervention modules for a 3-month
* Patients with no visit with Diabetes care provider within the 6 months prior to screening for study eligibility
* Pregnancy (only if subject, at the time of recruitment, reports being pregnant or planning a pregnancy in the next 6 months. Pregnancy tests will not be performed as part of the study).

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of interactive virtual educational module no. 1 | At completion of Module 1, at average of week 1
  Score on Likert-based scale on feedback survey.
Acceptability of interactive virtual educational module no. 2 | At completion of Module 2, at average of week 2
  Score on Likert-based scale on feedback survey.
Acceptability of interactive virtual educational module no. 3 | At completion of Module 3, at average of week 3
  Score on Likert-based scale on feedback survey.
Acceptability of interactive virtual educational module no. 4 | At completion of Module 4, at average of week 4
  Score on Likert-based scale on feedback survey.
Acceptability of interactive virtual educational module no. 5 | At completion of Module 5, at average of week 5
  Score on Likert-based scale on feedback survey.
Acceptability of interactive virtual educational module no. 6 | At completion of Module 6, at average of week 6
  Score on Likert-based scale on feedback survey.
Acceptability of interactive virtual educational module no. 7 | At completion of Module 7, at average of week 7
  Score on Likert-based scale on feedback survey.
Acceptability of interactive virtual educational module no. 8 | At completion of Module 8, at average of week 8
  Score on Likert-based scale on feedback survey.
Acceptability of interactive virtual educational module no. 9 | At completion of Module 9, at average of week 9
  Score on Likert-based scale on feedback survey.
Acceptability of interactive virtual educational module no. 10 | At completion of Module 10, at average of week 10
  Score on Likert-based scale on feedback survey.
Acceptability of interactive virtual educational module no. 11 | At completion of Module 11, at average of week 11
  Score on Likert-based scale on feedback survey.
Overall acceptability of entire interactive virtual educational program | At completion of Module 11, at average of week 11
  Score on Likert-based scale on feedback survey.
Attrition Rate | At completion of entire educational intervention for all participants, an average of 3-5 months
  Number of participants that did not complete the intervention divided by number of consenting participants
Recruitment Rate | At completion of recruitment of all participants, an average of 1 months
  Number of consenting participants divided by number of eligible approached candidates

SECONDARY OUTCOMES:
Change in subjective diabetes self-efficacy of participants | At baseline and at completion of entire educational intervention, an average of 3 months
  Comparison of pre and post intervention scores on Diabetes Empowerment Scale (Short form)- likert based scale
Change in participants' diabetes related knowledge | At baseline and at completion of entire educational intervention, an average of 3 months
  Comparison of pre and post intervention scores on Diabetes knowledge test (assessed through percent correct answers on an multiple choice test)
Change in participants' diabetes related distress | At baseline and at completion of entire educational intervention, an average of 3 months
  Comparison of pre and post intervention scores on likert based scale called Problem Areas in Diabetes Scale (for 20 to 21 years old participants) and Problem Areas in Diabetes- Teen Scale (for 16-19 years old participants).
Change in participants' Time In Range | At baseline and at completion of entire educational intervention, an average of 3 months
  Comparison of pre and post intervention Time in Range data from Continuous Glucose monitor.
Change in participants' HBA1C | At baseline and at completion of entire educational intervention, an average of 3 months
  Comparison of pre and post intervention HBA1C
Correlation of outcome expectation on degree of change in participants subjective diabetes self-efficacy after the educational intervention. | At completion of entire educational intervention, an average of 3 months
  Outcome Expectation evaluated with a survey consisting of 5 questions.
Correlation of outcome expectation on degree of change in participants diabetes related knowledge after the educational intervention. | At completion of entire educational intervention, an average of 3 months
  Outcome Expectation evaluated with a survey consisting of 5 questions.
Correlation of outcome expectation on degree of change in participants diabetes related distress after the educational intervention. | At completion of entire educational intervention, an average of 3 months
  Outcome Expectation evaluated with a survey consisting of 5 questions.
Correlation of outcome expectation on degree of change in participants HBA1C after the educational intervention. | At completion of entire educational intervention, an average of 3 months
  Outcome Expectation evaluated with a survey consisting of 5 questions.
Correlation of outcome expectation on degree of change in participants Time in Range after the educational intervention. | At completion of entire educational intervention, an average of 3 months
  Outcome Expectation evaluated with a survey consisting of 5 questions.

OTHER OUTCOMES:
Correlation of childhood opportunity index (COI) with degree of change in participants' subjective diabetes self-efficacy after the educational intervention. | At completion of entire educational intervention, an average of 3 months
  COI is measure of quality of resources and conditions for children's development (scale of 1-5, where 1 is worst COI and 5 is the best COI)
Correlation of childhood opportunity index (COI) with degree of change in participants' diabetes related knowledge after the educational intervention. | At completion of entire educational intervention, an average of 3 months
  COI is measure of quality of resources and conditions for children's development (scale of 1-5, where 1 is worst COI and 5 is the best COI)
Correlation of childhood opportunity index (COI) with degree of change in participants' diabetes related distress after the educational intervention. | At completion of entire educational intervention, an average of 3 months
  COI is measure of quality of resources and conditions for children's development (scale of 1-5, where 1 is worst COI and 5 is the best COI)
Correlation of childhood opportunity index (COI) with degree of change in participants' HBA1C after the educational intervention. | At completion of entire educational intervention, an average of 3 months
  COI is measure of quality of resources and conditions for children's development (scale of 1-5, where 1 is worst COI and 5 is the best COI)
Correlation of childhood opportunity index (COI) with degree of change in participants' Time In Range after the educational intervention. | At completion of entire educational intervention, an average of 3 months
  COI is measure of quality of resources and conditions for children's development (scale of 1-5, where 1 is worst COI and 5 is the best COI)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Wood, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nathan DM; DCCT/EDIC Research Group. The diabetes control and complications trial/epidemiology of diabetes interventions and complications study at 30 years: overview. Diabetes Care. 2014;37(1):9-16. doi: 10.2337/dc13-2112. PMID 24356592
- [Background] Mortensen HB, Hougaard P. Comparison of metabolic control in a cross-sectional study of 2,873 children and adolescents with IDDM from 18 countries. The Hvidore Study Group on Childhood Diabetes. Diabetes Care. 1997 May;20(5):714-20. doi: 10.2337/diacare.20.5.714. PMID 9135932
- [Background] Jack L. Biopsychosocial factors affecting metabolic control among female adolescents with type 1 diabetes. Diabetes Spectrum. 2003;16(3):154-159.
- [Background] Helgeson VS, Siminerio L, Escobar O, Becker D. Predictors of metabolic control among adolescents with diabetes: a 4-year longitudinal study. J Pediatr Psychol. 2009 Apr;34(3):254-70. doi: 10.1093/jpepsy/jsn079. Epub 2008 Jul 30. PMID 18667479
- [Background] Miller KM, Foster NC, Beck RW, Bergenstal RM, DuBose SN, DiMeglio LA, Maahs DM, Tamborlane WV; T1D Exchange Clinic Network. Current state of type 1 diabetes treatment in the U.S.: updated data from the T1D Exchange clinic registry. Diabetes Care. 2015 Jun;38(6):971-8. doi: 10.2337/dc15-0078. PMID 25998289
- [Background] Schilling LS, Knafl KA, Grey M. Changing patterns of self-management in youth with type I diabetes. J Pediatr Nurs. 2006 Dec;21(6):412-24. doi: 10.1016/j.pedn.2006.01.034. PMID 17101399
- [Background] Sigurdardottir AK. Self-care in diabetes: model of factors affecting self-care. J Clin Nurs. 2005 Mar;14(3):301-14. doi: 10.1111/j.1365-2702.2004.01043.x. PMID 15707440
- [Background] Tsang SK, Hui EK, Law BC. Self-efficacy as a positive youth development construct: a conceptual review. ScientificWorldJournal. 2012;2012:452327. doi: 10.1100/2012/452327. Epub 2012 Apr 29. PMID 22645423
- [Background] Winkley K, Ismail K, Landau S, Eisler I. Psychological interventions to improve glycaemic control in patients with type 1 diabetes: systematic review and meta-analysis of randomised controlled trials. BMJ. 2006 Jul 8;333(7558):65. doi: 10.1136/bmj.38874.652569.55. Epub 2006 Jun 27. PMID 16803942
- [Background] Hood KK, Rohan JM, Peterson CM, Drotar D. Interventions with adherence-promoting components in pediatric type 1 diabetes: meta-analysis of their impact on glycemic control. Diabetes Care. 2010 Jul;33(7):1658-64. doi: 10.2337/dc09-2268. PMID 20587726
- [Background] Viner RM, Christie D, Taylor V, Hey S. Motivational/solution-focused intervention improves HbA1c in adolescents with Type 1 diabetes: a pilot study. Diabet Med. 2003 Sep;20(9):739-42. doi: 10.1046/j.1464-5491.2003.00995.x. PMID 12925054
- [Background] Grey M, Boland EA, Davidson M, Li J, Tamborlane WV. Coping skills training for youth with diabetes mellitus has long-lasting effects on metabolic control and quality of life. J Pediatr. 2000 Jul;137(1):107-13. doi: 10.1067/mpd.2000.106568. PMID 10891831
- [Background] Laffel LM, Vangsness L, Connell A, Goebel-Fabbri A, Butler D, Anderson BJ. Impact of ambulatory, family-focused teamwork intervention on glycemic control in youth with type 1 diabetes. J Pediatr. 2003 Apr;142(4):409-16. doi: 10.1067/mpd.2003.138. PMID 12712059
- [Background] Nansel TR, Iannotti RJ, Simons-Morton BG, Cox C, Plotnick LP, Clark LM, Zeitzoff L. Diabetes personal trainer outcomes: short-term and 1-year outcomes of a diabetes personal trainer intervention among youth with type 1 diabetes. Diabetes Care. 2007 Oct;30(10):2471-7. doi: 10.2337/dc06-2621. Epub 2007 Jul 9. PMID 17620445
- [Background] Krishna G, Mathur JS, Gupta RK. Health hazard amongst chrome industry workers with special reference to nasal septum perforation. Indian J Med Res. 1976 Jun;64(6):866-72. No abstract available. PMID 977043
- [Background] Wood CL, Clements SA, McFann K, Slover R, Thomas JF, Wadwa RP. Use of Telemedicine to Improve Adherence to American Diabetes Association Standards in Pediatric Type 1 Diabetes. Diabetes Technol Ther. 2016 Jan;18(1):7-14. doi: 10.1089/dia.2015.0123. Epub 2015 Aug 21. PMID 26295939
- [Background] Guttmann-Bauman I, Kono J, Lin AL, Ramsey KL, Boston BA. Use of Telehealth Videoconferencing in Pediatric Type 1 Diabetes in Oregon. Telemed J E Health. 2018 Jan;24(1):86-88. doi: 10.1089/tmj.2017.0072. Epub 2017 Jun 27. PMID 28654350